CLINICAL TRIAL: NCT02238873
Title: Pegfilgrastim on Day +3 Compared to Day +1 for Patients With Refractory or Relapsed Aggressive Lymphoma Receiving Salvage Chemotherapy - a Randomized Controlled Trial
Brief Title: Pegfilgrastim on Day +3 Compared to Day +1 After Salvage Chemotherapy for Patients With Refractory or Relapsed Aggressive Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, LIAT VIDAL FISHER, MD MSc, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEGFIL
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Lymphoma; Neutropenia
Keywords: lymphoma; neutropenia; pegfilgrastim
MeSH Terms: conditions — Lymphoma; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegfilgrastim +1 (Active Comparator): Pegfilgrastim will be given 24 hours (day +1) after completion of salvage chemotherapy
  Interventions: Drug: Pegfilgrastim
- Pegfilgrastim +3 (Experimental): Pegfilgrastim will be given 72 hours (day +3) after completion of salvage chemotherapy
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim
  Other Names: Neulastim

SUMMARY:
Granulocyte colony stimulating factors (GCSFs) stimulate the level of white blood cells, specifically neutrophils. GCSF support for patients receiving chemotherapy was shown to decrease the rate of fever during low neutrophil count (neutropenia), and in some cancer types may decrease mortality. Pegfilgrastim is a pegylated form of the GCSF named filgrastim. Pegfilgrastim is used to stimulate bone marrow to produce more neutrophils to fight infection in patients undergoing chemotherapy. It has a much longer half-life than the parent filgrastim. It is removed from the body within the neutrophils. According to the American Society of Clinical Oncology 2006 guidelines pegfilgrastim should be given 24 hours after the completion of chemotherapy i.e.before neutrophil count starts to drop. Therefore it is cleared before and after neutropenia. Comparative low quality studies suggest that deferring pegfilgrastim delivery until neutrophil counts start dropping may result in improved its efficacy. This was further tested in a few small randomized controlled trials (high quality studies, considered the "gold standard" of studies) in different settings (including first chemotherapy for lymphoma, and solid cancer) with inconsistent results. Pegfilgrastim (given 24 hours after completion of chemotherapy) is a standard part of any salvage chemotherapy for patient with refractory or relapsed aggressive lymphoma. The investigators plan a randomized controlled trial comparing the efficacy of pegfilgrastim given 72 hours (day +3) vs. 24 hours (day +1) after completion of salvage chemotherapy in patients with refractory or relapsed aggressive lymphoma. The investigators will evaluate whether that change of pegfilgrastim schedule affects the risk of fever during neutropenia, neutrophil count, length of hospitalization, mortality, and safety.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age 18 years or above)

* Refractory or relapsed aggressive lymphoma, including Hodgkin's and non-Hodgkin's lymphoma
* Candidate for salvage chemotherapy. Salvage chemotherapy includes one of the following regimens: Ifosfamide, etoposide, vincristine (ICE), Cisplatin, cytarabine, and dexamethasone (DHAP), Etoposide, methylprednisolone, cytarabine, cisplatin (ESHAP). Chemotherapy dose reduction will be allowed.
* Chemotherapy with or without immunotherapy
* Therapy in hospital or at the outpatient clinic

Exclusion Criteria:

* Indolent lymphoma; we will exclude patients with transformed lymphoma.
* Treatment with GCSFs for the primary disease (e.g. aplastic anemia, MDS).
* Uncontrolled infection
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Febrile neutropenia | 30 days
  Number of participants with fever and neutropenia
Neutrophil count <500/ mcL | day 8 to 10
  Number of participants with neutrophil count below 500 /mcL

SECONDARY OUTCOMES:
Mortality | 30 days
  Number of participants who died by day 30
Neutrophil count <100/ mcL | day 8 to 10
  Number of patients with neutrophil count below 100/ mcL
Number of febrile days | 30 days
  a febrile day defined by at least one documented temperature measurement >38ºC
Development of clinically documented infections (CDI), microbiologically-documented infections (MDI) and clinically-significant bloodstream infections (BSI), not present at the time of randomization | 30 days
  Number of participants with CDI, MCI or BSI. CDI, MDI and BSI will be defined in accordance with the CDC surveillance definitions for healthcare-associated infections
Hospitalization | 30 days
  Number of hospitalization days of each participant (excluding days of hospitalization for chemotherapy)
Adverse events | 30 days
  ECOG common toxicity criteria grading Number of patients with an adverse event (AE). Number of patients with grade 3-4 AE

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel